CLINICAL TRIAL: NCT05534516
Title: Physiologic Changes Associated With Health Deterioration, Medications and Fluids Used in the Telemetry Unit
Brief Title: A Study of Physiologic Changes in a Telemetry Unit
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Antonio J. Forte, Principal Investigator, Mayo Clinic
Other Study IDs: 22-006064
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Acute Illness Requiring to Hospital Telemetry Admission

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the physiological changes associated with health deterioration, as well as different types, doses, and routes of administration of medications and fluids in acutely ill patients.

ELIGIBILITY:
Inclusion Criteria: Mayo Clinic patients who:

* Admitted to telemetry unit
* With acute illness
* Received any type of medication via any route of administration (oral, sublingual, intranasal, inhalational, intramuscular, intravenous, subcutaneous, transdermal)
* Received any amount of any type of intravenous fluids
* Cognitively and/or physically be able to sign consent

Exclusion Criteria:

- None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18-65 years) admitted to the telemetry unit at Mayo Clinic Florida's Hospital with acute illness followed from admission to discharge.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Rate | Baseline, through telemetry unit stay (approximately 1-3 days)
  Number of beats per minute
Change in Blood Pressure | Baseline, through telemetry unit stay (approximately 1-3 days)
  Measured in millimeters of mercury (mmHg)
Change in Respiratory Rate | Baseline, through telemetry unit stay (approximately 1-3 days)
  Number of breaths per minute
Change in Oxygen Saturation Levels | Baseline, through telemetry unit stay (approximately 1-3 days)
  Measured by a pulse oximeter reading reported as a percentage
Change in ECG morphology | Baseline, through telemetry unit stay (approximately 1-3 days)
  Changes in ECG waveform appearance measured from the digital ECG waveform interpretation

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Forte, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials